CLINICAL TRIAL: NCT01204775
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Saxagliptin (BMS-477118) as Monotherapy in Pediatric Patients With Type 2 Diabetes
Brief Title: Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Saxagliptin as Monotherapy in Pediatric Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV181-058; 2010-020360-38 (EudraCT Number)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxagliptin (Experimental): Saxagliptin Tablet, 2.5 mg, or Saxagliptin Tablet, 5 mg, (based on subject's weight)
  Interventions: Drug: Saxagliptin; Drug: Metformin (Active Rescue)
- Placebo (Placebo Comparator): Placebo matching saxagliptin tablet
  Interventions: Drug: Placebo (Saxagliptin); Drug: Metformin IR; Drug: Placebo (Metformin); Drug: Metformin (Active Rescue)

INTERVENTIONS:
Drug: Saxagliptin — Tablets, Oral, 2.5 mg or 5.0 mg (according to body weight category), Once Daily, 1-52 weeks
  Other Names: BMS-477118; Onglyza
  Arms: Saxagliptin
Drug: Placebo (Saxagliptin) — Tablets, Oral, Once daily, 1-16 weeks
  Arms: Placebo
Drug: Metformin IR — Tablets, Oral, 500 mg, Once Daily, 17-52 weeks
  Arms: Placebo
Drug: Placebo (Metformin) — Tablets, Oral, Once daily, 1-16 weeks
  Arms: Placebo
Drug: Metformin (Active Rescue) — Tablets, Oral, 500 mg, Titrated as needed, 2-52 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability, of Saxagliptin in pediatric patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients eligible if 10 years of age, up to 17 years and 32 weeks of age at the time of randomization, diagnosed as having type 2 diabetes prior to study enrollment.
* HbA1c ≥7.0% and ≤10.5%
* Body weight ≥ 30 kg.
* BMI > 85th percentile

Age and Reproductive Status a) Women of childbearing potential (WOCBP) and men must be using an acceptable method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized. The decision for appropriate methods to prevent pregnancy should be determined by discussions between the investigator and the study subject.

b) WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product. c) Women must not be breastfeeding. d) Sexually active fertile men must use effective birth control if their partners are WOCBP.

Exclusion Criteria:

1. Target Disease Exceptions

   a) Current use of the following medications for the treatment of diabetes, or use within the specified timeframe prior to screening for the study: i) Six months: insulin. ii) Four months: thiazolidinediones. iii) Two months: any other antidiabetic treatment iv) Any previous use of DPP4-inhibitor and/or incretin mimetics b) Current use of prescription or non-prescription weight loss drugs and their use within 3 months of screening.
2. Medical History and Concurrent Diseases

   a) Significant co-morbidity that, in the opinion of the investigators would preclude participation in the study (eg, current treatment for cancer). b) Previous diagnosis of monogenic etiology of type 2 diabetes such as MODY (maturity onset of diabetes in youth) or secondary diabetes (steroid use, Cushing's disease, acromegaly). c) Significant cardiovascular history. d) History of hemoglobinopathies (sickle cell anemia or thalassemias, sideroblastic anemia). e) History of unstable or rapidly progressive renal disease. f) History of alcohol or drug abuse. g) Psychiatric or cognitive disorder that will, in the opinion of investigators, limit the patient's ability to comply with the study medications and monitoring. h) Administration of any other study drug or participation in a clinical research trial within 30 days of planned enrollment to this study (or a longer period if dictated by local regulatory authorities). i) Any condition, which in the investigator's opinion may render the subject unable to complete the study or may pose significant risk to the subject. j) Immunocompromised individuals such as subjects that have undergone organ transplantation or subjects diagnosed with human immunodeficiency virus. k) Subjects on a commercial weight loss program with ongoing weight loss, or on an intensive exercise program.
3. Physical and Laboratory Test Findings a) Fasting plasma glucose (FPG) > 255 mg/dL (14.2 mmol/L) at screening will exclude the patient. b) Diabetic ketoacidosis (DKA) within 6 months of study entr1) Target Disease Exceptions a) Current use of the following medications : i) Six months: insulin. ii) Four months: thiazolidinediones. iii) Two months: any other antidiabetic treatment iv) Any previous use of DPP4-inhibitor and/or incretin mimetics b) Current use of prescription or non-prescription weight loss drugs and their use within 3 months of screening.

2) Medical History and Concurrent Diseases

a) Significant co-morbidity that, in the opinion of the investigators would preclude participation in the study (eg, current treatment for cancer). b) Previous diagnosis of monogenic etiology of type 2 diabetes such as MODY (maturity onset of diabetes in youth) or secondary diabetes (steroid use, Cushing's disease, acromegaly). c) Significant cardiovascular history. d) History of hemoglobinopathies (sickle cell anemia or thalassemias, sideroblastic anemia). e) History of unstable or rapidly progressive renal disease. f) History of alcohol or drug abuse. g) Psychiatric or cognitive disorder that will, in the opinion of investigators, limit the patient's ability to comply with the study medications and monitoring. h) Administration of any other study drug or participation in a clinical research trial within 30 days of planned enrollment to this study (or a longer period if dictated by local regulatory authorities). i) Any condition, which in the investigator's opinion may render the subject unable to complete the study or may pose significant risk to the subject. j) Immunocompromised individuals such as subjects that have undergone organ transplantation or subjects diagnosed with human immunodeficiency virus. k) Subjects on a commercial weight loss program with ongoing weight loss, or on an intensive exercise program. 3) Physical and Laboratory Test Findings

1. Fasting plasma glucose (FPG) > 255 mg/dL (14.2 mmol/L) at screening
2. Diabetic ketoacidosis (DKA) within 6 months of study entry (DKA can occur as a presenting sign of type 2 diabetes in youth).
3. Abnormal renal function, which is defined as an abnormal creatinine clearance rate as determined by the Schwartz Formula

Exclusion from study participation will apply to calculated glomerular filtration rate < 80 mL/min/1.73m2 (1.33 mL/s). d) Presence of one or more of the following: antibodies to glutamic acid decarboxylase (GAD), islet cell autoantibody (ICA), protein tyrosine phosphatase-like protein antibodies (IA-2). e) Active liver disease and/or significant abnormal liver function defined as Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2 times upper limits of normal, and/or serum total bilirubin > 2.0 mg/dL. f) History of positive serologic evidence of current infectious liver disease including anti-HAV (IgM), HbsAg, or anti-HCV. Patients who may have isolated positive anti HBs may be included. g) Anemia of any etiology defined as hemoglobin ≤ 10.7 g/dL (107 g/L) for females and ≤ 11.3 g/dL (113 g/L) for males. h) An abnormal TSH value at screening will be further evaluated by free T4. Subjects with an abnormal T4 will be excluded. i) Creatinine kinase (CK) ≥ 3 X ULN. j) Clinically significant (CS) abnormalities in any pre-randomization laboratory analyses or ECG that, in the investigator's opinion, would preclude randomization. 4) Allergies and Adverse Drug Reaction

1. Subjects who have contraindications to therapy as outlined in the Saxagliptin Investigator Brochure or local metformin package insert.
2. Subjects with known contraindications to DPP-IV therapy. 5) Prohibited Therapies and/or Medications

a) Steroid use exclusions: i) Excluded: use of oral or parenteral corticosteroids within 3 months ii) Allowed: inhaled corticosteroids for asthma, and topical corticosteroids if limited to minor surface area. b) Use of any other antihyperglycemic medication (other than metformin or insulin as applicable for glycemic rescue) after entry into the placebo lead-in period. c) Prior treatment with saxagliptin. d) Subjects taking prohibited medication as listed in Section 3.4. Subjects who stop prohibited medication prior to study participation must undergo an appropriate wash out period before visit 1. e) Diabetes treatment or use of weight loss medications f) Current treatment with potent CYP3A4/5 inhibitors (in countries where dose adjustment would be required by the saxagliptin label). 6) Sex and Reproductive Status

a) Pregnant, positive serum pregnancy test, planning to become pregnant during the clinical trials, or breastfeeding. 7) Other Exclusion Criteria

1. Prisoners or subjects who are involuntarily incarcerated.
2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
3. Employees of BMS, AstraZeneca (AZ), or their relatives.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2011-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (9):
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Hollywood, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Dearborn, Michigan
  - Research Site, Buffalo, New York
  - Research Site, Memphis, Tennessee
  - Research Site, Richmond, Virginia
- Russia (3):
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Pretoria
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 26 subjects enrolled, 12 subjects entered the lead in period. Of these 12 subjects, 8 subjects were randomized
Groups:
- Saxagliptin: Saxagliptin 2.5 mg or 5 mg depending on body weight
- Placebo: Placebo matching saxagliptin
Period: Overall Study
Arm/Group | Saxagliptin | Placebo
Started | 4 | 4
Double-blind Treatment Period | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1
Not completed — Poor/non-compliance | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in HbA1c From Baseline to Week 16
Time Frame: 16 week short term treatment period
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 4
percentage | -0.7 (0.83) | 0.6 (1.53)

ADVERSE EVENTS:
Time Frame: 52 week
Description: 16 week double-blind treatment period and 36 week long-term extension period
Arm/Group | Placebo | Saxagliptin
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Saxagliptin (N=4)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | Saxagliptin (N=4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
ACNE (Skin and subcutaneous tissue disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 1
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
VISION BLURRED (Eye disorders) | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0
PERIPHERAL SWELLING (General disorders) | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No